CLINICAL TRIAL: NCT01466556
Title: The Incidence of Metabolic Syndrome Among Obese Children in Our Region
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 80-2010-HYMC
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obese children
  Interventions: Other: Routine laboratory tests

INTERVENTIONS:
Other: Routine laboratory tests — Laboratory tests to determine metabolic syndrome

SUMMARY:
The aim of this study is to determine the prevalence of metabolic syndrome amongst obese children in our region with a body mass index (BMI) above the 95th percentile for age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Children with BMI over 95 percentile

Exclusion Criteria:

* Obesity secondary to medication use
* Obesity secondary to genetic disease

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who visit our outpatient clinic or a routine visit to the ER
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of children with metabolic syndrome | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel